CLINICAL TRIAL: NCT00064467
Title: An 8 Week, Multicenter, Randomized, Double-blind, Placebo Controlled Comparison of the Efficacy of Extended Release Bupropion Hydrochloride and Placebo in the Treatment of Adult Outpatients With Major Depressive Disorder With Lethargic Symptoms
Brief Title: Lethargic Depression Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130931
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy; Major Depressive Disorder (MDD)
Keywords: lethargic; decreased interest; decreased motivation; depression
MeSH Terms: conditions — Epilepsy; Depressive Disorder, Major; Stupor; Depression

INTERVENTIONS:
Drug: Extended-release bupropion (HCl)

SUMMARY:
This is a study of Major Depressive Disorder (MDD) in patients with decreased energy, pleasure and interests.

DETAILED DESCRIPTION:
A Multicenter, Double-Blind, Placebo-controlled comparison of the efficacy and safety of flexible dose extended-release bupropion (HCl) 300-450 mg/day and placebo administered for eight weeks for the treatment of adult outpatients with major depressive disorder including symptoms of decreased energy, pleasure, and interest

ELIGIBILITY:
Inclusion criteria:

* Primary diagnosis of MDD with current duration lasting 12 weeks but no greater than 2 years.
* Generally in good health.
* Subject must read and write at a level sufficient to provide written informed consent.

Exclusion criteria:

* Current or past history of seizure disorder.
* Subject has a primary diagnosis or received treatment for panic disorder, obsessive compulsive disorder (OCD), post traumatic stress disorder (PTSD), acute stress disorder, Bipolar I or II disorder, schizophrenia, or other psychotic disorder.
* Currently using illicit drugs or other psychotropic drugs.
* Patient poses a current suicidal risk or has attempted suicide in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268
Dates: Start 2003-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from randomization on the Inventory of Depressive Symptomatology, self report and clinician rated.

SECONDARY OUTCOMES:
Percent of responders. Percent of remitters. Quality of Life Enjoyment and Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (24):
- United States (24):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Cromwell, Connecticut
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Middletown, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Ridgeland, Mississippi
  - GSK Investigational Site, Moorestown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, San Antonio, Texas

REFERENCES:
- [Result] Rush J, VanMeter SA, Wightman D, Hampton KD, Krishen A, Modell JG. Wellbutrin XL for the treatment of adults with major depressive disorder. American Psychiatric Association 158th Annual Meeting, Atlanta, GA, 21-26 May, 2005, Abstract No. 787.
- [Result] Jefferson JW, Rush AJ, Nelson JC, VanMeter SA, Krishen A, Hampton KD, Wightman DS, Modell JG. Extended-release bupropion for patients with major depressive disorder presenting with symptoms of reduced energy, pleasure, and interest: findings from a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2006 Jun;67(6):865-73. doi: 10.4088/jcp.v67n0602. PMID 16848645
- [Result] Rush J, VanMeter SA, Wightman DS, Hampton KD, Krishen A, Modell JG. Bupropion XL for the treatment of adults with major depressive disorder. 45th Annual New Clinical Drug Evaluation Unit (NCDEU) Meeting, Boca Raton, FL, 6-9June, 2005.